CLINICAL TRIAL: NCT03300934
Title: Adolescence and Diabetes: Can an Automated Closed Loop System Improve Control ?
Brief Title: Adolescence and Diabetes:Can an Automated Closed Loop System Improve Control ?
Acronym: SPIDIMAN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Luxembourg (Other)
Collaborators: University of Cambridge (Other); Luxembourg Institute of Health (Other Government)
Responsible Party: Principal Investigator, Carine de Beaufort, Guest professor, Centre Hospitalier du Luxembourg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Spidiman
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Type1 Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- closed loop glucose control system (Experimental): Closed loop glucose control system
  Interventions: Device: closed loop glucose control system
- CSII Pump treatment (No Intervention): CSII Pump treatment without the integrated algorithm and glucose sensor

INTERVENTIONS:
Device: closed loop glucose control system — Cross over between Closed loop glucose system with DANA pump, Navigator II CGM and Cambridge AP algorithm FD2A, versus usual CSII pump treatment
  Arms: closed loop glucose control system

SUMMARY:
This study evaluates the use of the FD2 automated closed loop insulin administration in Adolescents with a poor metabolic control . All youth will be treated in a random order by their usual pump treatment or an Automated system and we will evaluate whether this has an impact on metabolic control and sleep

DETAILED DESCRIPTION:
Achievement of a good metabolic control is very important for all persons with diabetes . In adolescence many changes occur , physically , socially and psychologically .This may influence the metabolic control . This study will evaluate whether the automated closed-loop will facilitate and improve the management of diabetes in youth with a poor metabolic control.

It is a single-centre, randomised, two-period crossover study to assess the efficacy /safety and acceptability of the automated closed-loop glucose control (CL) day and night, over 28 days in comparison with continuous subcutaneous insulin infusion (CSII) in the home setting in poorly controlled type 1 diabetes adolescents.

ELIGIBILITY:
Inclusion Criteria:

12- 18 years Type 1 diabetes according to WHO/ISPAD , for at least 1 year CSII treatment for at least 6 month HbA1c ≥ 8,0%, for more than 6 months Informed consent of the patient and parents

Exclusion Criteria:

Non-type 1 diabetes mellitus including those secondary to chronic disease Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator.

Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator Known or suspected allergy against insulin Recurrent incidents of severe hypoglycaemia as defined by ISPAD guidelines during the previous 12 months.

More than one episode of diabetic ketoacidosis (DKA) as defined by ISPAD in preceding 12 months

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Time spent in glucose target (%) (3.9 - 10 mmol/l) | 4 week treatment arms
  Continuous blinded glucose monitoring during the study period with and without the automated Closed loop on a between arm comparison.

SECONDARY OUTCOMES:
Time spent below glucose target (%) (<3.0mmol/l and < 2,5 mmol/l) | 4 week treatment arms
  Continuous blinded glucose monitoring during the study period with and without automated closed loop (%)
Time spent above glucose target (%) (> 10 mmol/l) | 4 week treatment arms
  Continuous blinded glucose monitoring during the study period with and without automated closed loop (%)
Severe hypoglycaemic events | 4 week treatment arms
  ISPAD Definition of severe hypoglycemia
Severe Diabetes ketoacidosis | 4 week treatment arms
  ISPAD definition of severe DKA
Use of the automated closed loop system (% time) | 4 week treatment arm
  % time , the system is used
Use of the CGM during closed loop | 4 week treatment arm
  % time , the system is used
Quality of life perception in adolescents | 4 week treatment periods
  Questionnaire based
Family Responsibility perception | 4 week treatment periods
  Questionnaire based : Family responsibility scale
User experience after the 4 week treatment | 4 week intervention
  questionnaire based

CONTACTS AND LOCATIONS:
Overall Officials: Carine de Beaufort, MD PhD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (1):
- Clinique des Enfants CHluxembourg, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No